CLINICAL TRIAL: NCT05635916
Title: A Prospective, Randomized Trial of Liposomal Bupivacaine Compared to Conventional Bupivacaine on Pain Control and Post-Operative Opioid Use in Receiving Adductor Canal Blocks for Total Knee Arthroplasty
Brief Title: Trial of Liposomal Bupivacaine for TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Light Mercy Hospital (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 155
Record Dates: First submitted 2022-09-26; First posted 2022-12-02 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Knee Replacement; Total Knee Arthroplasty; Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The randomization scheme will be developed using NQuery Software (Statistical Solutions, Boston, MA). The analyst will provide the research coordinator with randomization assignments in sequentially-numbered opaque envelopes. As the study is unblinded, both patients and providers will be aware of the randomization assignment. To help mitigate bias, the team members collecting and entering data will be masked regarding the patient's assignment. The REDCap database has the randomization assignments in an instrument separate from the study data collection instruments, allowing for data entry without seeing which group the subject is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine (Experimental): Adductor canal block using liposomal bupivacaine and conventional bupivacaine
  Interventions: Drug: Liposomal bupivacaine
- Standard of Care (Active Comparator): Adductor canal block using conventional bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Adductor canal block with injection of 10cc 13.3% liposomal bupivacaine combined with 10cc 0.50% bupivacaine within one hour following surgery
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine — Adductor canal block with injection of 20cc 0.5% bupivacaine within one hour following surgery
  Arms: Standard of Care

SUMMARY:
Total knee arthroplasty (TKA), also known as a knee replacement, is a procedure performed to reduce severe pain and improve function of the joint. Managing postoperative pain can be challenging following TKA, and inadequate relief can lead to impaired mobility and persistent opioid use. Adductor canal nerve blocks (ACB), have shown significant benefit in improving postoperative analgesia and patient satisfaction. However, the local anesthetic used currently for these blocks only provides temporary relief that wears off within 24 hours. Liposomal bupivacaine is an extended-release local anesthetic agent that can provide up to 72 hours of pain relief, however it is unclear if its use is also effective in ACBs for knee surgery. The purpose of this study is to determine if liposomal bupivacaine is better than conventional bupivacaine in improving pain control, opioid consumption, and length of stay in patients scheduled for TKA.

DETAILED DESCRIPTION:
BACKGROUND The femoral nerve block and the adductor canal nerve block are two regional anesthesia techniques used to manage pain control following TKA Femoral nerve blocks were the first peripheral nerve block employed for post-surgical analgesia, however they are now less frequently used due to significant drawbacks that influence recovery. The femoral nerve provides motor and sensory innervation to the quadriceps muscle. Blockade of the motor branches of this nerve leads to quadriceps weakness and increased risk of falling after surgery. Additionally, for similar reasons, ambulation after surgery can be significantly delayed. In contrast, the adductor canal block does not affect the quadriceps muscle, as it avoids the motor branches of the femoral nerve. The location of the block, located in the mid-thigh, mainly affects the sensory neuronal branches of the saphenous nerve. It has been found as a superior method for post-surgical analgesia since motor weakness is spared.

The adductor canal block is an interfascial plane block that can be performed as a single injection, or as a continuous infusion via insertion of a catheter. Continuous peripheral nerve blocks can provide prolonged post-operative analgesia, however, they are associated with several complications including catheter infection, obstructions, and fluid leakage Catheter placement takes a significant amount of time to perform and can consume valuable clinical resources. Additionally, catheter displacement can be frequent with ACBs, since the aponeurosis where the saphenous nerve lies is superficial, leading to easy dislodgement and block failure. In comparison, a single injection of local anesthetic in the adductor canal space is much simpler to place, is more cost effective, and has a lower infection risk. However, risk of rebound pain is much higher in single injection nerve blocks due to their shorter duration of action.

Liposomal bupivacaine (LB) is an extended-release local anesthetic that combines the benefits of a single injection nerve block with the long-lasting effects of continuous catheter infusions. LB received Food and Drug Administration approval in October 2011 for post-surgical anesthesia via local infiltration and, in April 2018, for interscalene brachial plexus blocks. LB has been reported to provide analgesia for up to 72 hours, making it the longest lasting local anesthetic currently available.

There have been several studies evaluating the effectiveness of perineural LB in improving peripheral nerve block analgesia compared to non-liposomal anesthetics for total knee arthroplasty but the evidence is not definitive. A meta-analysis performed found that LB was associated with higher pain relief compared to traditional bupivacaine and reduced opioid related complications in TKA patients. Another study found decreased opioid consumption and improved pain scores within the early post-operative period following TKA, but there was no significant difference in length of hospital stay, patient satisfaction, or adverse postoperative events. Another study found patients receiving LB for TKA had no improvement in narcotic use, length of stay, patient reported pain, or functional ability compared to those who received a single shot short acting ropivacaine nerve block. A recent meta-analysis concluded that perineural infiltration of LB in various, distinct peripheral nerve block locations was not superior to non-liposomal bupivacaine.

There is an institutional desire to improve postoperative pain outcomes and shorten length of stay in patients undergoing TKA. It is possible that liposomal bupivacaine may help improve these measures, however, current evidence is inconclusive. The purpose of this study is to investigate the analgesic efficacy of liposomal bupivacaine comparative to conventional bupivacaine in ACBs for individuals undergoing TKA.

SPECIFIC AIMS AND OVERALL SIGNIFICANCE Through this prospective trial, we aim to gather institutional data investigating the effectiveness of liposomal bupivacaine compared to conventional bupivacaine for the management of post-total knee arthroplasty pain.

Specific Aims Aim 1: To compare the efficacy of liposomal bupivacaine to conventional bupivacaine for adductor canal blocks in adults scheduled for total knee arthroplasty.

Aim 2: To compare postoperative opioid consumption measured as morphine milligram equivalents (MME) at 24 hours postoperatively.

Aim 3: To compare postoperative pain scores and opioid consumption at 48 and 72 hours after surgery.

Aim 4: To compare total length of postoperative stay following surgical stop time.

Significance This study is significant because there is conflicting evidence regarding the efficacy of liposomal bupivacaine. Currently, liposomal bupivacaine is used routinely at our institution for surgical wound infiltration. Liposomal bupivacaine is also routinely used at our institution for targeted peripheral nerve blocks for shoulder surgery.

Total knee arthroplasty is one of the most common surgeries performed to relieve joint pain in those suffering from arthritis of the knee.1 TKA is a procedure met with moderate to severe post-operative pain that affects early ambulation, range of motion, post-operative rehabilitation, patient satisfaction, and patient outcomes.1 Identifying optimal strategies to decrease acute pain is crucial for improving post-surgical outcomes in these patients. Although, similar to liposomal bupivacaine, continuous perineural catheters (PNC) can potentially provide greater than 24 hours pain relief while single shot nerve blocks with conventional local anesthetics typically provide less than 24 hours of pain relief, there are many factors which can impair PNC efficacy and their routine use for adductor canal blocks has fallen out of favor in recent years. Catheter placement can be quite challenging which can lead to block failure. Also, catheters can become dislodged, leak at the insertion site, and commonly get disconnected from the local anesthetic infusion pump, leading to interruption of analgesia. Since PNCs are an inserted foreign body, they carry a risk of infection greater than single shot local anesthetic techniques. Identifying an easy, reliable approach to provide multi-day pain relief will benefit patient care as well as current procedural and postoperative care workflows.

If our study reveals that liposomal bupivacaine can provide superior analgesia to standard single injection bupivacaine, this can have a profound impact on the future of post-TKA pain management.

MATERIALS AND METHODS This is a prospective, randomized, clinical trial comparing adductor canal blocks using liposomal bupivacaine to conventional bupivacaine for patients scheduled for total knee arthroplasty. Patients enrolled in this study will include those that are 18 years or older undergoing primary total knee arthroplasty and ASA class I-III. Patients that will be excluded are those that are unable to cooperate or consent to the study, have allergies to local anesthetics, have an infection at the needle insertion site, BMI >40 kg/m2, history of coagulopathy, substance use disorder diagnosis, and patients using opioids with greater than 90 MME/day.

STUDY PROTOCOL On the day of surgery, the anesthesiologist will elicit and answer any questions or concerns regarding the study. Patients will be informed of the potential risks and complications of nerve block placement that are inherent to their scheduled anesthetic and independent of their participation in the study. These include bleeding, infection, and potential nerve injury. Informed consent will be obtained from patients who were introduced to the study prior to the day of surgery and decide to enroll in the study.

After informed consent is obtained, patients will be randomized into the two study groups in a 1:1 ratio as follows:

Intervention arm: Adductor canal block with injection of 10cc 13.3% liposomal bupivacaine combined with 10cc 0.25% bupivacaine within one hour following surgery Control arm: Adductor canal block with injection of 20cc 0.5% bupivacaine within one hour following surgery (current standard practice) The randomization scheme will be developed using NQuery Software (Statistical Solutions, Boston, MA). The analyst will provide the research coordinator with randomization assignments in sequentially-numbered opaque envelopes. As the study is unblinded, both patients and providers will be aware of the randomization assignment. To help mitigate bias, the team members collecting and entering data will be masked regarding the patient's assignment. The REDCap database has the randomization assignments in an instrument separate from the study data collection instruments, allowing for data entry without seeing which group the subject is in.

The ultrasound guided nerve blocks will be performed by experienced study staff members of the regional anesthesia team. Patients will be placed on standard ASA monitors and given supplemental O2 via nasal cannula or simple mask. The injection site(s) will be prepped and draped using standard infection control and sterile protocols. Light sedation will be given as needed by the attending anesthesiologist, and skin infiltration of the puncture site with 2% lidocaine will be performed.

An ultrasound will be used to visualize the saphenous nerve and any relevant structures. After the targeted nerve structures have been identified, the peripheral nerve block needle will be advanced under direct ultrasound visualization. Following negative aspiration of blood and air, the study drug will be deposited in the immediate vicinity of the saphenous nerve using low pressure injections.

In the event of poorly controlled pain at any point during the study, we will provide the patient with appropriate analgesic rescue agents to ensure that post-surgical pain is adequately controlled. All pain medications will be documented for subsequent analysis.

Outcome data will be collected by a blinded member of the anesthesia research team as outlined in the data collection table. Vital signs, NRS pain scores, and adverse symptoms will be recorded in the subject's medical record as standard practice. This information will be collected for study purposes.

If a participant decides to withdraw from the study prior to the 72 hour time point, data collected prior to withdrawal will be included in the study unless the subject requests that their data be removed from the study database.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older who are scheduled for a total knee arthroplasty at Northern Light Mercy Hospital

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of liposomal bupivacaine to conventional bupivacaine for adductor canal blocks in adults scheduled for total knee arthroplasty. | Measured at 24 hours post-op
  The primary outcome of this study will be composite pain scores 24 hours after surgery. Others have shown that composite pain scores quantify pain with greater accuracy than a single measurement. Jensen et. al. concluded in their study that composite pain intensity scores from two or more individual ratings of pain are valid for detecting treatment effects.23 Pain scores will be measured using a numeric rating scale (NRS) (0=no pain; 10= worst possible pain) "Worst," "average," and "least" pain scores will be assessed for the preceding time interval at 24, 48, and 72 hours following surgery. If a participant is discharged prior to 72 hours after surgery, they will be given a log to record their pain scores and pain medication use to report to study staff via telephone.
To compare postoperative pain scores and opioid consumption at 48 hours after surgery. | Measured at 48 hours post-op
  The primary outcome of this study will be composite pain scores 24 hours after surgery. Others have shown that composite pain scores quantify pain with greater accuracy than a single measurement. Jensen et. al. concluded in their study that composite pain intensity scores from two or more individual ratings of pain are valid for detecting treatment effects.23 Pain scores will be measured using a numeric rating scale (NRS) (0=no pain; 10= worst possible pain) "Worst," "average," and "least" pain scores will be assessed for the preceding time interval at 24, 48, and 72 hours following surgery. If a participant is discharged prior to 72 hours after surgery, they will be given a log to record their pain scores and pain medication use to report to study staff via telephone.
To compare postoperative pain scores and opioid consumption at 72 hours after surgery. | Measure at 72 hours post-op
  The primary outcome of this study will be composite pain scores 24 hours after surgery. Others have shown that composite pain scores quantify pain with greater accuracy than a single measurement. Jensen et. al. concluded in their study that composite pain intensity scores from two or more individual ratings of pain are valid for detecting treatment effects.23 Pain scores will be measured using a numeric rating scale (NRS) (0=no pain; 10= worst possible pain) "Worst," "average," and "least" pain scores will be assessed for the preceding time interval at 24, 48, and 72 hours following surgery. If a participant is discharged prior to 72 hours after surgery, they will be given a log to record their pain scores and pain medication use to report to study staff via telephone.

SECONDARY OUTCOMES:
To compare postoperative opioid consumption measured as morphine milligram equivalents (MME) at 24 hours postoperatively. | Measured intraoperatively, in PACU at 4 hours post-op, and at 24,48, and 72 hours post-op.
  For our opioid consumption assessments, data will be collected intraoperatively, in the PACU at 4 hours post-op, and at the 24hr, 48hr, and 72hr timepoints following surgery, as is standard for surgical patients. Information on opioid type and dose will be obtained through review of the participant's electronic medical record or through phone assessment, depending on point of hospital discharge. Opioid amounts will be converted into MMEs.
To compare total length of postoperative stay following surgical stop time. | Measure at discharge, an average of 1 day.
  The time of surgical stop time and discharge will be extracted from the medical record and calculated to length of stay in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Brian McAllister, MD, Principal Investigator — Medical Staff & Chief of Anesthesia
Locations (1):
- Northern Light Mercy Hospital, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quaye A, McAllister B, Garcia JR, Nohr O, Laduzenski SJ, Mack L, Kerr CR, Kerr DA, Razafindralay CN, Richard JM, Craig WY, Rodrigue S. A prospective, randomized trial of liposomal bupivacaine compared to conventional bupivacaine on pain control and postoperative opioid use in adults receiving adductor canal blocks for total knee arthroplasty. Arthroplasty. 2024 Feb 1;6(1):6. doi: 10.1186/s42836-023-00226-y. PMID 38297390